CLINICAL TRIAL: NCT00278005
Title: Incidence of Infection in the Patient With DiGeorge Syndrome Following Surgery for Congenital Heart Disease
Brief Title: Infection in DiGeorge Following CHD Surgery
Status: Terminated | Type: Observational
Why Stopped: completed
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 05-134
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2008-03

CONDITIONS: DiGeorge Syndrome; Congenital Heart Defects
Keywords: pediatric; DiGeorge Syndrome; Congenital heart defects; Infections; Cardiac surgery
MeSH Terms: conditions — DiGeorge Syndrome; Heart Defects, Congenital; Infections

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We propose a retrospective review of patients with DiGeorge syndrome having undergone cardiac surgery to evaluate the incidence of blood stream and/or surgical site infection. The hypothesis is that we will find an increased number of infections for this sub-group. We will compare the incidence of infection to children of similar age and diagnosis to evaluate for variances in the incidence of infection.

DETAILED DESCRIPTION:
DiGeorge syndrome is a common genetic disorder that frequently results in congenital heart defects such as truncus arteriousus, coarctation of the aorta, interrupted aortic arch, tetralogy of Fallot, pulmonary atresia with VSD, and several others. The defect is usually due to a deletion in the long arm of chromosome 22. Approximately 25% of patients with DiGeorge have a congenital heart defect. These patients also have varying degrees of thymic hypoplasia with associated T cell dysfunction. They are at increased risk of infections and can be at risk for opportunistic infections when the degree of T cell dysfunction is severe. Children undergoing cardiac surgery are at risk for infections in the post-operative period, prolonging hospital stay and increasing morbidity and mortality. The patient with DiGeorge syndrome may have higher rates of infection due to associated immune system dysfunction, however, this has not been previously reported from a large group of DiGeorge syndrome patients. Children's Healthcare of Atlanta follows over 200 patients with DiGeorge syndrome, with the majority having previously undergone cardiac surgery. This group of patients may benefit from more extensive antibiotic prophylaxis following surgery if they indeed have significantly higher rates of infection, but the true incidence needs to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Children's Healthcare of Atlanta patients, Egleston DiGeorge Syndrome Cardiac Surgery 200 medical charts between Jan 1, 1998 and April 31, 2005 with cardiac surgery and DiGeorge Syndrome 200 medical charts between Jan 1, 1998 and April 31,2005 with cardiac surgery and no DiGeorge Syndrome

Exclusion Criteria:

* Those who do not meet inclusion criteria

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: DiGeorge Syndrome Cardiac Surgery
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 1998-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O Maher, MD, Principal Investigator — Children's Healthcare of Atlanta, Sibley Heart Center Cardiology
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States